CLINICAL TRIAL: NCT04800887
Title: Comparison of Visual Outcomes and Contrast Sensitivity in Patients Implanted With Tecnis Eyhance IOL (Intraocular) and Tecnis Monofocal IOL
Brief Title: Visual Outcomes and Contrast Sensitivity in Patients Implanted With Tecnis Eyhance Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Andrea Janekova, MD, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEY-VAO
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Intraocular Lens
Keywords: EDOF lens; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: each patient in group received monofocal intraocular lens in one eye and extended depth of focus intraocular lens in second eye
Who Masked: Participant, Investigator
Masking Description: Double masked- patient and investigator are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended depth of focus intraocular lens (Active Comparator): Eyes of patients implanted with extended depth of focus lens Tecnis Eyhance
  Interventions: Device: TECNIS Eyhance intraocular lens
- Monofocal intraocular lens (Active Comparator): Eyes of patients implanted with monofocal lens Tecnis ZCB00
  Interventions: Device: Monofocal intraocular lens Tecnis ZCB00

INTERVENTIONS:
Device: TECNIS Eyhance intraocular lens — Cataract surgery and implantation with extended depth of focus intraocular lens
  Arms: Extended depth of focus intraocular lens
Device: Monofocal intraocular lens Tecnis ZCB00 — Cataract surgery and implantation with monofocal intraocular lens
  Arms: Monofocal intraocular lens

SUMMARY:
To compare visual outcomes for various distances, reading speed, contrast sensitivity, glare occurence, defocus curve and subjective satisfaction in patients implanted with the extended depth of focus lens (Tecnis Eyhance) in one eye and monocal aspheric lens (Tecnis ZCB00) in second eye. Patients undergo visit in 3,6 and 12 months after the surgery.

DETAILED DESCRIPTION:
The goal of refractive cataract surgery is to remove the opacity, or cataract and to produce the desired refractive outcome. In most cases, the desired outcome is an emmetropic eye, or an eye that sees 20/20 Snellen for distance vision post-surgery with the implant of a monofocal IOL. This, however, does not offer much in the way of intermediate and near vision. The increased desire for simultaneous distance, intermediate and near vision has increased the popularity of multifocal IOLs (MIOLs). However MIOLs provide visual acuity for all distances, they has occurence of optical phenomena such as glare and halo and lower contrast sensitivity. Extended depth of focus (EDOF) lens should provide distance vision as good as monofocal lens and intermediate vision better than monofocal but without any optical phenomenon or decreased contrast sensitivity.

This study is conducted from 11/2019 to 08/2021 in the Ophthalmology department of Faculty Hospital Kralovske Vinohrady in Prague. The research protocol was explained to all participants and informed consent was signed before enrolling patient to the study. The study was approved by the Ethics Committee of Faculty Hospital Kralovske Vinohrady and will enrolled up to 25 patients with presence of cataract in both eyes.

Bilateral clear corneal phacoemulsification and IOL implantation is performed by one surgeon using the same technique in both eyes. The surgical process involved topical anesthesia, superior 3-step clear corneal incision (2,2mm), 5,0mm curvilinear capsulorhexis, phacoemulsification, bilateral irrigation- aspiration and IOL implantation. One eye is implanted with EDOF IOL second eye with monofocal IOL. Type of IOL is chosen randomly and double masked.

Patients are scheduled for visit at 3,6 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* presence of cataract in both eyes
* no other ocular pathology affecting visual acuity
* bilateral phacoemulsification cataract surgery was arranged for both eyes
* corneal astigmatism up to 0,75 cylinder (measured by IOL Master biometry)
* dioptric power of both selective lens within 1,5 D range in one patient
* selecting IOL power between 18 D and 27 D power range

Exclusion Criteria:

* complicated cataract
* corneal opacities or irregularities
* amblyopia
* anisometropia
* coexisting ocular pathologies
* glaucoma
* history of ocular surgery
* refusal or unable to maintain follow-up

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Comparison of visual acuity between eyes implanted with EDOF IOL and eyes implanted with monofocal IOL | 12 months
  * uncorrected distance visual acuity (UDVA)
  * corrected distance visual acuity (CDVA)
  * uncorrected near visual acuity (UNVA)
  * distance corrected near visual acuity (DCNVA)
  * corrected near visual acuity (CNVA)
  * uncorrected intermediate visual acuity (UIVA)
  * distance corrected intermediate visual acuity (DCIVA)
Comparison of reading speed between eyes implanted with EDOF IOL and eyes implanted with monofocal IOL | 12 months
  Monocular reading speed (Salzburg reading desk for 66cm and 80cm)
Difference in contrast sensitivity between eyes with EDOF IOL and monofocal IOL | 12 months
  Contrast sensitivity - CSV (contrast sensitivity vision) 1000 device- monocularly, mesopic, without glare Contrast sensitivity measurement on Glaretester- monocularly- with and without glare
Comparison of defocus curve between eyes implanted with EDOF IOL and eyes implanted with monofocal IOL | 6 months
  A defocus curve that measures visual acuity should be obtained by using the best corrected distance refraction and then defocusing the image in 0.5 increments from +1.5 to -2.5 diopter with spherical plus and spherical minus trial lenses (i.e.,+1.5 D, +1.0 D, +0.5 D, 0.00 D, -0.5 D, -1.00 D, . . . ,-2.50 D) with visual acuity recorded at each change in correction.

SECONDARY OUTCOMES:
Questionaire | 6 months
  Questionaire based on Catquest-9SF (9-item short-form) questionaire with special questions of feeling difference in vision in each eye for various distances Contains questions for activities for various distances with scale of difficulty of doing activity without glasses from 1-4 (1= Yes, very great difficulty, 4= No, no difficulty and Cannot decide answer).
  Contains more 3 questions for feeling difference in visual acuity between eyes.
Change in intermediate visual acuity in eyes implanted with EDOF IOL | 3 and 12 months
  * uncorrected intermediate visual acuity (UIVA) - photopic condition
  * distance corrected intermediate visual acuity (DCIVA)- photopic condition
Change in reading speed in eyes implanted with EDOF IOL | 3 and 12 months
  Salzburg reading desk for 66cm and 80cm
Change in contrast sensitivity in eyes implanted with EDOF IOL | 3 and 12 months
  Contrast sensitivity - CSV (contrast sensitivity vision) 1000 device- mesopic, without glare Contrast sensitivity measurement on Glaretester - with and without glare

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Janekova, MD, Principal Investigator — Faculty Hospital Kralovske Vinohrady
Locations (1):
- Faculty hospital Kralovske Vinohrady, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No